CLINICAL TRIAL: NCT06771596
Title: A Prospective, Single-arm Study on Nimotuzumab Combined With Concurrent Chemoradiotherapy for the Treatment of Locally Advanced High-risk Squamous Cell Carcinoma of the Cervix
Brief Title: Nimotuzumab High-risk, Locally Advanced Squamous Cell Carcinoma of the Cervix
Acronym: CC11
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SHUANG ZHENG JIA, PhD, Attending Physician, Ph. D., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-IST-CC-20210304; Y-QL202101-0108 (Other Grant/Funding Number: CSCO-Qilu Cancer Research Fund)
Record Dates: First submitted 2024-12-28; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Uterine Cervical Neoplasms
Keywords: nimotuzumab; high-risk locally advanced cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemoradiotherapy + nimotuzumab (Experimental): Participants receive nimotuzumab 400 mg intravenously (IV) on Day 1 of each week cycle (QW) for 4-6 cycles . During the period of nimotuzumab, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 4- 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy .The cumulative dose at Point A/HRCTV D90 should be equal to or greater than 87 Gy EQD2Gy. The combination of brachytherapy and external beam radiotherapy should be completed within 8 weeks.
  Interventions: Drug: Nimotuzumab Injection

INTERVENTIONS:
Drug: Nimotuzumab Injection — Nimotuzumab is a highly humanized monoclonal antibody of IgG1 type, with a humanization rate of 95%. It is highly specific, has a long half - life, and shows high selectivity and a high degree of humanization. It can specifically block the epidermal growth factor receptor (EGFR) signaling pathway and mediate immune effects such as antibody - dependent cell - mediated cytotoxicity (ADCC) and complement - dependent cytotoxicity (CDC). It also promotes the endocytosis and degradation of EGFR, thereby inhibiting the proliferation of tumor cells and promoting the apoptosis of tumor cells, reversing the malignant biological behavior of tumor cells at the molecular level.
  Other Names: Nimotuzumab

SUMMARY:
The efficacy and safety of nimotuzumab in the treatment of high-risk, locally advanced squamous cell carcinoma of the cervix.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of nimotuzumab plus concurrent chemoradiotherapy in the treatment of high-risk locally advanced cervical squamous cell carcinoma.

This study adopts a single-arm design, and the primary efficacy endpoint is the 2-year progression-free survival (PFS) rate.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old.
* Newly diagnosed cervical squamous cell carcinoma confirmed by histology, with a clinical stage of stage III - IVA (FIGO 2018 staging).
* No prior receipt of surgery, radiotherapy, or systemic anticancer therapy for the treatment of cervical cancer.
* No previous exposure to the study drug.
* Presence of at least one measurable or evaluable lesion as per RECIST version 1.1, with the measurable lesion exhibiting a longest diameter of ≥10 mm on spiral CT scan or a shortest diameter of ≥15 mm for enlarged lymph nodes, which has not been previously irradiated.
* Absence of central nervous system diseases, both primary and metastatic.
* WHO/ECOG performance status score of 0-1.
* Anticipated survival duration of at least 12 weeks.
* Adequate organ function within the following parameters (without the use of any blood components, cytokines, or growth factors within 14 days prior to randomization):

  1. Absolute neutrophil count (ANC) ≥1.5×10^9/L
  2. Platelet count ≥90×10^9/L
  3. Hemoglobin level ≥90 g/L
  4. Serum albumin level ≥30 g/L
  5. Bilirubin level ≤1.5 times the upper limit of normal (ULN)
  6. Alanine transaminase (ALT) and aspartate transaminase (AST) levels ≤3×ULN
  7. Serum creatinine level ≤1.5×ULN
  8. Thyroid-stimulating hormone (TSH) level ≤1×ULN (with eligibility also extended to patients with free triiodothyronine [FT3] or free thyroxine [FT4] levels ≤1×ULN).
* For women of childbearing potential not undergoing surgical sterilization, a negative serum pregnancy test (hCG) within 72 hours prior to study randomization is required; breastfeeding must be absent. Additionally, the use of a medically approved contraceptive method is mandatory from the time of informed consent through the study treatment period and for 120 days following the final administration of the trial medication or 180 days after the last chemotherapy/ radiotherapy session. Participants must also agree not to donate eggs for reproductive purposes or to freeze/preserve eggs for this use during the aforementioned period.
* Informed consent must be obtained with documentation.
* Availability for follow-up assessments.

Exclusion Criteria:

* Cervical adenocarcinoma and other rare pathological types.
* Having previously received surgical treatment, pelvic radiotherapy, systemic chemotherapy, tumor targeted therapy, or immunotherapy for cervical cancer.
* Bilateral hydronephrosis, unless resolved by unilateral stent placement or percutaneous nephrostomy, or deemed mild and without clinical significance by the investigator.
* Pregnant women or those in the lactation period.
* With rectovaginal fistula/vaginal vesical fistula/uncontrolled massive vaginal bleeding or at risk of developing a fistula.
* Active infectious processes necessitating antimicrobial therapy, including the use of antibacterial, antiviral, or antifungal agents.
* History of immunodeficiency, including HIV seropositivity or other acquired and congenital immunodeficiency disorders.
* Uncontrolled cardiac symptoms or diseases, such as NYHA class II or higher heart failure, unstable angina, myocardial infarction within the past year, atrial fibrillation, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, PR interval greater than 250 ms, or QTc interval ≥470 ms.
* History of other malignant tumors (except for cured basal cell carcinoma of the skin).
* Crohn's disease or ulcerative colitis.
* Allergic to nimotuzumab or its components.
* contraindications for cisplatin use.
* Neurological or mental disorders affecting cognitive ability.
* Unable to receive intracavitary radiotherapy.
* Other reasons not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | 24 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD.

SECONDARY OUTCOMES:
Overall Survival (OS) at Month 24 | 24 months
  OS is the time from randomization to death due to any cause. OS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the OS rate at Month 24 using the entire OS data up to the cut-off date.
Complete Response Rate | 3-6 months
  Complete response refers to the situation where, after treatment, all target lesions (in the evaluation of cancer treatment, these are the tumor sites that are predetermined for observing and assessing the curative effect) completely disappear, no new lesions emerge, and the tumor markers (if there are relevant markers for evaluating the disease) return to normal levels. The complete response rate refers to the proportion of patients who have achieved a complete response state among all the patient groups receiving treatment.
Objective Response Rate | 3-6 months
  The Objective Response Rate (ORR) is an important indicator for measuring the effectiveness of cancer treatment. It refers to the proportion of patients whose tumors shrink to a predefined value and can maintain it for the minimum time requirement. Specifically, it includes patients with complete response (CR) and partial response (PR). As mentioned before, complete response means that all target lesions completely disappear, no new lesions appear, and the relevant tumor markers are normal. Partial response refers to the situation where the product of the maximum diameter and its maximum perpendicular diameter of a single tumor lesion (for a single lesion) or the sum of the maximum diameters of all target lesions (for multiple lesions) shrinks by a certain proportion (usually more than 30%), while no new lesions appear and there is no progression of non-target lesions.
Disease Control Rate | 3-6 months
  The Disease Control Rate (DCR) is a crucial indicator for evaluating the effectiveness of cancer treatment. It refers to the proportion of patients whose tumors achieve complete response (CR), partial response (PR), and stable disease (SD) among the total number of patients after treatment. Stable disease means that the product of the maximum diameter and its maximum perpendicular diameter of a single tumor lesion (for a single lesion) or the sum of the maximum diameters of all target lesions (for multiple lesions) neither shrinks to an extent sufficient to be judged as partial response nor enlarges to an extent sufficient to be judged as progressive disease (PD), and at the same time, no new lesions appear.
Duration of Response | 24 months
  The duration of response refers to the time interval starting from the time when the tumor was first recorded to meet the response criteria (complete response, CR or partial response, PR), and ending at the time when the tumor was first found to have progressive disease (PD) or when death occurred due to any reason.
Time to Progression | 24 months
  Time to Progression (TTP) refers to the time from when a patient starts receiving treatment to when the tumor shows progressive disease (PD).
Number of Participants Who Experience One or More Adverse Events | 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shuangzheng Jia, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China